CLINICAL TRIAL: NCT01756560
Title: A Study of the Effect of Dexamethasone on Duration of Lower Extremity Blocks With Bupivacaine in Subjects Having ACL Repair
Brief Title: Effect of Dexamethasone on Duration of Lower Extremity Blocks With Bupivacaine in Subjects Having ACL Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to continue research due to time constraints
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB12-2191
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Duration of Pain Relief
Keywords: anterior cruciate ligament; block duration
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): in this group, plain bupivacaine will be used to block femoral and sciatic nerve
  Interventions: Drug: Bupivacaine
- Dexamethasone (Experimental): Bupivacaine mixed with dexamethasone will be used to block femoral and sciatic nerve
  Interventions: Drug: dexamethsone; Drug: Bupivacaine

INTERVENTIONS:
Drug: dexamethsone
  Arms: Dexamethasone
Drug: Bupivacaine

SUMMARY:
Anterior cruciate ligament reapair is a painful procedure. Single shot femoral and sciatic nerve block only last 12-16 hrs. Since dexamethasone prolongs brachial plexus block, using it in lower extremity blocks will prolong the analgesia to provide better outpatient pain relief after surgery at home.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75, no contraindication to regional anesthesia

Exclusion Criteria:

* peripheral neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Malik, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: in this group, plain bupivacaine will be used to block femoral and sciatic nerve
  Bupivacaine
- Dexamethasone: Bupivacaine mixed with dexamethasone will be used to block femoral and sciatic nerve
  dexamethsone
  Bupivacaine
Period: Overall Study
Arm/Group | Control | Dexamethasone
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: study terminated prematurely
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Dexamethasone | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Analgesia Duration
Time Frame: 72 hours
Population: study terminated early due to lack of resources to recruit subjects and no data was collected for Outcome measures
Arm/Group | Control | Dexamethasone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No